CLINICAL TRIAL: NCT01546233
Title: Outcome of Multidisciplinary Education Programme in Self-care in Fatigue Lung Cancer Patients Who Receiving Chemotherapy Treatment
Brief Title: Multidisciplinary Education in Lung Cancer Patients Who Receiving Chemotherapy Treatment
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: RajavithiMultidisciplinary01
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Chemotherapy; Multidisciplinary self care programme; Fatigue
MeSH Terms: conditions — Lung Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- multidisiplinary self care program: Patient with Lung cancer will be participated in group education with multidisiplinary self care program
  Interventions: Behavioral: multidisciplinary education programme
- Conventional education: Lung cancer patient will be received standard education
  Interventions: Behavioral: standard education

INTERVENTIONS:
Behavioral: multidisciplinary education programme — Educate of self-care by Oncology nurses to relieve and prevent the fatigue of cancer chemotherapy, and provide the manual to read at home, take about 15 minutes. By using home exercise program, 30 minutes of physical education. Teaching and demonstration exercises of the muscles to breath and conservation of energy during exercise and record the exercise/walking diary, the nutritional education nutrition counseling, psychiatric assessment,self-care prevention of depression.
  Other Names: multidisciplinary self care education programm
  Groups: multidisiplinary self care program
Behavioral: standard education — standard education before and after chemotherapy
  Other Names: standard education before and after chemotherapy
  Groups: Conventional education

SUMMARY:
The purpose of this study is to compare the fatigue in lung cancer patients receiving chemotherapy treatment, between the education programme in self-care a multidisciplinary with the group who received standard care.

DETAILED DESCRIPTION:
Educate of self-care by Oncology nurses to relieve and prevent the fatigue of cancer chemotherapy, and provide the manual to read at home, take about 15 minutes. By using home exercise program, 30 minutes of physical education. Teaching and demonstration exercises of the muscles to breath and conservation of energy during exercise and record the exercise/walking diary, the nutritional education nutrition counseling, psychiatric assessment,self-care prevention of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 45-65 years.
2. Has been diagnosed lung cancer stages 3-4 must be chemotherapy is platinum-based, and had received chemotherapy for at least one time, must be in the range of 2-4 cycles of chemotherapy.
3. Performance status: ECOG 0-1
4. No problem hearing it.
5. Read and write Thai.
6. Be willing to cooperate in research. And signed a joint research

Exclusion Criteria:

1. The complications include: high fever, severe nausea and vomiting.
2. Injection drug use in diabetes treatment.
3. Ischemic heart disease with heart arrhythmia and the drug continuously.
4. Is unable to daily living. Caused by defects in movement, and severe osteoarthritis, muscle atrophy, paralysis or walking flat less than 10 meters.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fatigue Lung Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measure fatigue by questionnaires | August 2011 to august 2012 (up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Kotchukorn Wnagnum, Msc (nurse), Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Department of Chemotherapy Unit, Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
๋Journal of the medical association of Thailand